CLINICAL TRIAL: NCT05729360
Title: "An Open Safety Study and Description of the Parameters of the Therapeutic Efficacy of the Drug for Early Etiotropic Therapy for Coronavirus Infection Caused by the SARS-CoV-2 Virus, With a Single Application in Patients With Confirmed COVID-19 Diagnosis"
Brief Title: Study of Monoclonal Antibodies for Early Etiotropic Therapy for Coronavirus Infection Caused by the SARS-CoV-2 Virus
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Gamaleya Research Institute of Epidemiology and Microbiology, Health Ministry of the Russian Federation (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 02-GamCoviMab-2022
Record Dates: First submitted 2023-02-06; First posted 2023-02-15 (Actual); Last update posted 2023-02-15 (Actual); Status verified 2023-02

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients with a verified diagnosis of COVID-19 (Experimental)
  Interventions: Drug: GamCoviMab

INTERVENTIONS:
Drug: GamCoviMab — A total of 30 people will be randomized and receive the study drug (GamCoviMab) in a hospital setting (7 days of hospitalization).

SUMMARY:
Open prospective non-comparative study of safety and tolerability of the drug (GamCoviMab) with the description of the parameters of the therapeutic efficacy in patients with confirmed COVID-19 diagnosis.

ELIGIBILITY:
Inclusion Criteria:

Each potential patient for inclusion in the study must meet all of the following criteria:

1. Presence of a written Informed Consent to participate in the study;
2. Men and women aged 18 to 75 years inclusive;
3. Positive SARS-CoV-2 test result ≤5 days prior to enrollment or clinical manifestations later confirmed by PCR;
4. Oxygen saturation ≥93% without oxygen donation by any means, diagnosed with COVID-19 disease with symptom onset within 5 days of inclusion;
5. Presence of several symptoms of mild or moderate severity at the time of inclusion in the study;
6. At the time of screening for the study, the patient is not hospitalized;
7. Presence of high risk factors for severe COVID-19 and/or hospitalization and/or death, in the opinion of the investigator, not limited to the following:

   1. not fully vaccinated and unvaccinated patients
   2. elderly patients (over 60), including those with additional risk factors
   3. obesity
   4. immunocompromised patients, including those receiving immunosuppressive drugs for any indication
   5. with comorbidities (diabetes, diseases of the cardiovascular system, coagulopathy, chronic kidney disease, including conditions requiring dialysis, chronic lung disease, liver disease, etc.)
8. Consent to use effective methods of contraception during the entire period of participation in the study.
9. Able to carry out study visits.

Exclusion Criteria:

The patient will not be included in the study in the following cases:

1. Inability to read Russian; inability or unwillingness to understand the essence of the study. Any other condition that limits the eligibility of obtaining informed consent or may affect the volunteer's ability to participate in the study;
2. Pregnancy or breast-feeding;
3. Severe and extremely severe course of COVID-19:

   * Oxygen saturation at rest according to pulse oximetry (SpO2) ≤ 93% OR
   * PaO2/FiO2 ≤ 300 mm Hg OR
   * Respiratory failure and need for invasive mechanical ventilation (with tracheal intubation) or ECMO OR
   * Septic shock OR
   * Multiple organ failure
4. Prior therapy with plasma from a recovered COVID-19 patient or other anti-SARS CoV-2 mAbs for the treatment of current COVID-19 disease at study entry;
5. The patient is currently hospitalized or, in the opinion of the investigator, may require hospitalization within the next 24 hours;
6. Requires oxygen therapy due to COVID-19 disease or requires an increase in basal oxygen flow due to COVID-19 disease in individuals on chronic oxygen therapy due to non-COVID-19 related comorbidities;
7. Confirmed active tuberculosis, AIDS;
8. The presence of any life-threatening decompensated comorbidity which, in the opinion of the Investigator, makes the patient unsuitable for inclusion in the study;
9. Body weight less than 40 kg;
10. Volunteer participation in any other clinical trial within the last 90 days;
11. Requires mechanical ventilation or the inevitable need for mechanical ventilation in the next 24 hours based on the current state of the patient;
12. Suspected or proven serious active bacterial, fungal, viral, or other infection (other than COVID-19) that, in the opinion of the investigator, may pose a risk to the volunteer and affect the assessment of study endpoints;
13. There are concomitant diseases requiring surgical intervention within the next month;
14. Aggravated allergic history (including, but not limited to, erythema multiforme major, toxic epidermal necrolysis, Quincke's edema, polymorphic exudative eczema, a history of serum sickness, hypersensitivity or allergic reactions to the administration of immunobiological drugs, known allergic reactions to drug components, etc.);
15. Severe infusion reactions in history;
16. Alcohol or drug addiction.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-03 (Estimated); Primary Completion 2023-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Occurrence of adverse events (AE) | within 28 days after administration of the drug
  Occurrence of adverse events (AE) within 28 days after administration of the drug
Occurrence of serious adverse events (SAEs) | within 180 days after administration of the drug
  Occurrence of serious adverse events (SAEs) throughout the study